CLINICAL TRIAL: NCT06115902
Title: A Phase 1 Clinical Trial of TQB2102 for Injection in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) -Expressing Relapsed/Metastatic Breast Cancer
Brief Title: A Study of TQB2102 for Injection in Patients With Recurrent/Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-Ib-01
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2102 for injection (Experimental): Dose: 6.0 mg/kg or 7.5 mg/kg of TQB2102 for injection. Administration: Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle.
  Interventions: Drug: TQB2102 for injection

INTERVENTIONS:
Drug: TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC)

SUMMARY:
TQB2102 is an antibody-drug conjugate comprised of a humanised antibody against Human Epidermal Growth Factor Receptor 2 (HER2), an enzyme-cleavable linker, and a topoisomerase I inhibitor payload, which combine the ability of antibodies to specifically target tumour cells with the highly potent killing activity of drugs with payloads too toxic for systemic administration. This is a Phase 1/Phase 2 study to evaluate the effectiveness, safety, pharmacokinetics (PK) and anti-drug antibody (ADA) of TQB2102 for injection in subjects with HER2-expressing relapsed/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Between the ages of 18-75 years (subject to the date of signing the informed consent); Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥3 months;
* Breast cancer patients diagnosed with HER2 expression by pathological examination, with evidence of local focal recurrence or distant metastasis, are not suitable for surgery or radiotherapy for cure;
* Disease progression or intolerance during or after the most recent treatment period must be present before participating in clinical trials;
* At least one measurable lesion (based on Response Evaluation Criteria In Solid Tumors 1.1);
* The main organs function are normally;
* Female participants of childbearing age should agree to use contraception during the study period and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male participants should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Concomitant disease and medical history:

  1. Has diagnosed and/or treated additional malignancy within 3 years prior to first administration of study drug;
  2. Adverse effects due to any prior treatment have not been restored according to CommonTerminology Criteria for Adverse Events (CTCAE) 5.0 ≤ level 1 (Excluding hair loss);
  3. Major surgical treatment, incision biopsy, or significant traumatic injury received within 28 days prior to study treatment;
  4. Long-term unhealed wounds or fractures;
  5. Patients who have a prior history of interstitial lung disease/pneumonia requiring steroid intervention, or who are present with interstitial lung disease/pneumonia, or who are suspected of having interstitial lung disease/pneumonia on screening imaging and cannot be ruled out;
  6. Arterial/venous thrombosis events, such as cerebrovascular accident, deep vein thrombosis, and pulmonary embolism, occurred within 6 months before the first medication;
  7. Patients who have a history of psychotropic substance abuse and are unable to abstain or have mental disorders;
  8. Patients with any severe and/or uncontrolled disease;
* Tumor related symptoms and treatment:

  1. Patients who have been treated with other antitumor drug, such as chemotherapy, radical radiotherapy, or immunotherapy, within 4 weeks prior to the first dose, or who are still within 5 half-lives of the drug;
  2. Received Chinese patent drugs with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions within 2 week before the study treatment;
  3. Patients whose imaging shows that the tumor has invaded important blood vessels or who are determined by the investigators to be highly likely to invade important blood vessels during follow-up studies and cause fatal major bleeding;
  4. Uncontrolled pleural effusion, ascites, and moderate or higher pericardial effusion requiring repeated drainage;
  5. Known presence of cancerous meningitis or clinically active central nervous system metastasis; Patients who have been stable for at least 4 weeks after treatment and have been off corticosteroids for at least 2 weeks are excluded;
  6. Patients with severe bone injury due to tumor bone metastasis;
* Study treatment related: people who are known to be allergic to the study drug or its excipients, or to humanized monoclonal antibody products;
* Patients who participated in and used other anti-tumor clinical trials within 4 weeks before the first medication;
* In the judgment of the investigator, there is a situation that seriously endangers the safety of the subjects or affects the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 10 months.
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Baseline up to 14 months.
  PFS defined as the time from the first injection until the first documented progressive disease (PD) or death from any cause, whichever happens first.
Duration of Remission (DOR) | Baseline up to 14 months.
  DOR defined as the time when the participants first achieved complete or partial remission to disease progression.
Disease Control Rate (DCR) | Baseline up to 10 months.
  Percentage of participants achieving complete response (CR), partial response (PR) and stable disease (SD).
Clinical Benefit Rate (CBR) | Baseline up to 14 months.
  Percentage of participants achieving complete response (CR), partial response (PR) and stable disease (SD) for ≥ 24 weeks.
Overall Survival (OS) | Baseline up to 20 months.
  OS defined as the time from the first injection to death from any cause.
Incidence of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The occurrence of all adverse medical events after the first injection.
Severity of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The severity of all adverse medical events after the first injection.
Concentration of TQB2102 | 0 to 1 hour before infusion and 0.5 to 2 hours after infusion on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1 and Cycle 7 Day 1. Each cycle is 21 days.
  Serum concentration of TQB2102
Concentration of total antibody | 0 to 1 hour before infusion and 0.5 to 2 hours after infusion on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1 and Cycle 7 Day 1. Each cycle is 21 days.
  Total antibody concentration in serum
Small molecule toxin | 0 to 1 hour before infusion and 0.5 to 2 hours after infusion on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1 and Cycle 7 Day 1. Each cycle is 21 days.
  Small molecule toxin in plasma
Anti-drug antibody (ADA) | Before infusion on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, Cycle 12 Day 1, 30 days after the end of the last infusion. Each cycle is 21 days.
  Incidence of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Anhui Pronvincial Cancer Hospital, Hefei, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University School of Medicine, Xi'an, Shannxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang